CLINICAL TRIAL: NCT06463314
Title: A Prospective Cross-Sectional Study to Evaluate Performance and Usability of Multiplo® TP/HIV Test at Point-Of-Care Sites in the Hands of Untrained Non-Health Care Professional Operators
Brief Title: Multiplo Near Patient Non-HCP Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The device manufacturer is no longer seeking licensure for this use-case in Canada.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REACH Multiplo TP/HIV-01
Record Dates: First submitted 2024-05-31; First posted 2024-06-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections; Syphilis Infection
Keywords: point of care; health care provider; screen test; device trial
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: screening for HIV and syphilis infection at point of care settings by untrained non-professional health care providers
Masking Description: blinded study design involving participants with known and unknown syphilis and HIV status where test providers are blinded to the participant status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants with known and unknown HIV and/or syphilis status (Experimental): All participants will undergo fingerstick blood testing with the test device administered by untrained non-professional health care providers, along with venous blood testing at a central laboratory using licensed gold standard comparator methods.
  Interventions: Device: Multiplo TP/HIV Antibody Test

INTERVENTIONS:
Device: Multiplo TP/HIV Antibody Test — The Multiplo TP/HIV Antibody Test (MedMira Laboratories Inc., Halifax, NS), ["Multiplo TP/HIV Test"] is a single use, rapid, vertical-flow in vitro qualitative immunoassay for the detection of antibodies to Human Immunodeficiency Virus (HIV) Type 1/Type 2 and Treponema pallidum (Syphilis) in human fingerstick blood. The Multiplo® TP/HIV Test is intended as an aid in the diagnosis of HIV1/2 and Syphilis infections in patients with signs and symptoms of HIV and syphilis. The test is intended for use by trained personnel in medical facilities, clinical laboratories, emergency care situations, and physicians' offices as an in vitro diagnostic device capable of providing results in less than five minutes. The Multiplo TP/HIV Test has not yet sought approval for self-testing. All required pre and post-test counselling guidelines must be followed in each setting in which the Multiplo TP/HIV Test is used. Results are read visually.

SUMMARY:
To help reach the undiagnosed living with HIV and/or syphilis in Canada, point-of-care (POC) tests for HIV and Syphilis may have substantial utility for increased identification of infected individuals through their relative ease of use and portability, as well as their ability to deliver rapid, actionable results while the care provider still has access to the patient. MedMira Inc. (Halifax, NS, Canada), has developed a POC test to detect HIV and Syphilis antibodies in fingerstick blood samples that is seeking approval from Health Canada for use by trained healthcare professionals. The goal of this study is to provide evidence that untrained, non-registered health care providers (ie. peer testers) can perform the test without any increased risk of obtaining erroneous results. This test requires no instrumentation and can be used by non-registered health care professionals including peer testers ("Operators") in multiple near patient settings such as community health centres and point of care testing locations.

DETAILED DESCRIPTION:
This is a blinded, controlled study to evaluate the ability of the Operators, including peer testers, to perform and interpret the HIV and Syphilis results of the Multiplo TP/HIV Test. The non-registered health care professionals including peer testers are defined as non-health care professional (ie. Peers) paid site personnel that have no training or hands-on experience with the Multiplo Test. This protocol involves collection of fingerstick whole blood from a minimum of 800 Participants to test with the Multiplo Test. Testing will be conducted by the study Operators in near-patient clinical settings. Results from the Multiplo Test will be compared to results from blood based serological assays, including licensed 4th generation HIV EIA and syphilis EIA/RPR assays. Study Operator qualifications and assessment of the ease of device use will be evaluated. Operators will also read and interpret various contrived devices in order to assess their ability to correctly interpret a variety of potential test results.

All enrolled Participants will voluntarily provide medical history and the specimens according to Section 4, Study Procedures at Visit 1 (Day 1), for the testing with the Multiplo Test.

All Participants will have a laboratory test done for performance comparison, but only those with unknown HIV and/or syphilis status will be instructed to return to the clinic for a follow-up visit (Visit 2), two (2) weeks later to obtain their laboratory test results. Participants may also have a separate Point-of-Care (POC) test for HIV and/or syphilis conducted on site as part of the clinic's standard of care testing, outside of the protocol.

Activities in the plan of the study include:

* Selection of study Operators with informed consent for participation in the study
* Completion of Untrained Operator Eligibility and Assessment Questionnaire - prior to study start
* Screening of participants and obtaining informed consent
* Review of inclusion/exclusion criteria and completion of Participant Enrollment Questionnaire
* Specimen Collection and Testing:

  * Collection of venous blood for Clinical Laboratory testing for HIV and Syphilis
  * Collection of fingerstick whole blood for testing with the Multiplo Test
* Laboratory testing for HIV and Syphilis
* Clinical follow up for Participants with positive HIV and/or Syphilis test results from Clinical Laboratory testing
* Participants who test negative will have opportunities for preventative services including PrEP
* Completion of Untrained Operator Usability and Interpretation Questionnaire - after study completion
* Untrained non-professional Operator Mock Device Interpretation Assessment Following recruitment of participants and obtaining informed consent, Participants may be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria

Participants considered eligible for inclusion are those who:

* Are at least 18 years of age
* Are able to read/understand English or French
* Are able to provide informed consent
* Agree to provide accurate medical history
* Are able to provide up to 20mL blood by venipuncture, and a small amount of blood by fingerstick
* Agree to undergo testing for HIV and syphilis with the Multiplo® TP/HIV Test
* For the Participants previously diagnosed with HIV and/or syphilis, diagnosis can have occurred at any time prior to enrolment
* For the Participants with negative or unknown HIV and/or syphilis status - last HIV negative test must be greater than 3 months prior to date of consent

Exclusion Criteria

Participants considered ineligible for participation in the trial are those who meet any of the following exclusion criteria:

* Are site employees
* Are in the judgment of the investigator to be unable to complete the study or are unlikely to comply with the study protocol
* Have been previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent positive and negative agreement of the Multiplo® TP/HIV Test performed by non-healthcare providers to the Participant's HIV and/or syphilis status confirmed by the lab results. | 6 months
  The primary outcome for the study will be the percent positive and negative agreement of the Multiplo® TP/HIV Test performed by intended, untrained users to the Participant's HIV and/or syphilis status confirmed by the lab results. The percentages for positive and negative agreement will be calculated with the two-sided 95% confidence intervals for both as follows: % Positive Agreement= ((n) HIV or syphilis Multiplo reactive results )/((n) HIV or syphilis positive status)×100 % Negative Agreement= ((n)HIV or syphilis Multiplo non reactive results )/((n) HIV or syphilis negative status)×100 Percent positive and negative agreement will be calculated for each analyte (HIV or syphilis) separately.

SECONDARY OUTCOMES:
Percent of correctly interpreted mock devices by untrained, non-healthcare professional operators | 6 months
  Non-health care professionals will be asked to read results from a variety of mock test results. These mock tests will be blind coded, provided to the non-HCP in random order followed by review and documentation of the panels of contrived test results to be interpreted by study Operators. The results indicated by the non-HCP will be compared against the code to determine the ability of the non-HCP to correctly interpret a variety of results including, strong positive, weak positive, invalid, weak negative and strong negative. will be given a panel of

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Cool Aid Community Health Centre, Victoria, British Columbia
  - Nine Circles Community Health Centre, Winnipeg, Manitoba
  - Hassle Free Clinic, Toronto, Ontario
  - Women's Health in Women's Hands, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660